CLINICAL TRIAL: NCT02660333
Title: Effect of Prebiotic or Synbiotic Supplementation on Inflammatory Response and Indicators of Nutritional Status in Individuals With Morbid Obesity: A Randomized Clinical Trial, Placebo-controlled and Triple Blind
Brief Title: Effect of Prebiotic or Synbiotic on Inflammatory Response and Indicators of Nutritional Status in Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Catarina (Other)
Responsible Party: Principal Investigator, Erasmo Benicio Santos de Moraes Trindade, Doctor, Universidade Federal de Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UFSC
Record Dates: First submitted 2016-01-14; First posted 2016-01-21 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Morbid Obesity
Keywords: Obesity; Inflammation; Nutritional status; Prebiotic; Synbiotic
MeSH Terms: conditions — Obesity, Morbid; Obesity; Inflammation | interventions — Prebiotics; Synbiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study participants and researchers were masked over consumption and distribution of supplementation, respectively. Laboratory technicians who performed the blood collection were also masked as to the distribution of supplementation. Supplements and placebo were pre-packaged by the supplier in opaque and closed sachets with randomization codes, being identical in physical appearance, taste and color. Supplement identification codes were only disclosed by the supplier after statistical analysis of study data.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Placebo
- Prebiotic (Active Comparator): Fructooligosaccharide
  Interventions: Dietary Supplement: Prebiotic
- Synbiotic (Active Comparator): Fructooligosaccharide + Lactobacillus paracasei LPC-37 + Lactobacillus rhamnosus HN001 + Lactobacillus acidophilus NCFM + Bifidobacterium lactis HN019
  Interventions: Dietary Supplement: Synbiotic

INTERVENTIONS:
Dietary Supplement: Placebo — Maltodextrin - 11g/day
  Arms: Placebo
Dietary Supplement: Prebiotic — Fructooligosaccharide - 11g/day
  Arms: Prebiotic
Dietary Supplement: Synbiotic — Fructooligosaccharide + Lactobacillus paracasei LPC-37 + Lactobacillus rhamnosus HN001 + Lactobacillus acidophilus NCFM + Bifidobacterium lactis HN019 - 11g/day
  Arms: Synbiotic

SUMMARY:
The purpose of this study is to evaluate the effect of prebiotic or synbiotic supplementation on inflammatory response and indicators of nutritional status in patients with morbid obesity. Study hypothesis: Supplementation of 12 g/day of fructooligosaccharides (prebiotic) or 12 g/day of fructooligosaccharides + strains of lactobacilli and bifidobacteria (synbiotic) during 30 days promotes reduction of plasma/serum levels of acute phase proteins, cytokines, metabolic and anthropometric parameters in individuals with BMI ≥ 40kg/m².

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of prebiotic or synbiotic supplementation on inflammatory response and indicators of nutritional status in patients with morbid obesity. Adult individuals of both sexes with morbid obesity (body mass index ≥ 40 kg/m²) will be invited to participate in this randomized, placebo-controlled, triple-blind study. The participants will be divided into three groups: G1 - control group (placebo), G2 - prebiotic group and G3 - synbiotic group. The study will consist of four experimental time points: M0 - baseline and start of supplementation; M1 - after fifteen days of the first outpatient visit and fifteen days after the start of supplementation with prebiotic, synbiotic or placebo; M2 - after thirty days from the first outpatient visit and end of supplementation with prebiotic, synbiotic and placebo; and M3 - time after sixty days from the first outpatient visit. At all time points the inflammatory response will be assessed by determination of plasma cytokines (IL-1, IL-6, IL-10, TNF) and acute phase proteins (c-reactive protein and albumin), besides the evaluation of laboratory and anthropometric indicators of nutritional status. The primary endpoint will be the reduction in concentrations of inflammatory markers (cytokines and acute phase proteins).

Investigators expect to contribute with new information in this field of knowledge, which may facilitate the clinical application of these results.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years and less than 60 years
* Body mass index (BMI)≥40kg/m2

Exclusion Criteria:

* Previous gastrointestinal diseases (e.g. cancer and inflammatory bowel disease)
* Intolerances and/or food allergies (e.g. lactose intolerance and celiac disease)
* Current use of anti-inflammatory drugs and/or antibiotics and/or immunosuppressants
* Regular use of laxatives and/or appetite suppressants
* Current or previous use (up to one month) of prebiotics, probiotics, synbiotics or products enriched with these food compounds
* Intolerance to prebiotic and/or probiotic and/or synbiotic
* Following a diet for weight loss in the last three months
* Pregnant or breastfeeding
* Following unusual diets (e.g. vegetarian, macrobiotic)
* Alcohol dependence and/or illicit drugs dependence
* Smokers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
C-reactive protein | 2 months
  Serum C-reactive protein concentrations (mg/L)
Cytokines | 2 months
  Plasma IL-1, IL-6, IL-8, IL-10, IL-12p70 and TNF-alpha concentrations (pg/mL)

SECONDARY OUTCOMES:
Triglycerides | 2 months
  Serum concentrations of triglycerides (mg/dL)
Total cholesterol | 2 months
  Serum concentrations of total cholesterol (mg/dL)
LDL-c | 2 months
  Serum concentrations of LDL-cholesterol (mg/dL)
HDL-c | 2 months
  Serum concentrations of HDL-cholesterol (mg/dL)
Blood glucose | 2 months
  Blood glucose concentrations (mg/dL)
Glycated hemoglobin | 2 months
  Blood concentrations of glycated hemoglobin (%)
Growth hormone | 2 months
  Serum concentrations of Growth hormone (ng/mL)
Fasting insulin | 2 months
  Serum concentrations of insulin (IU/mL)
Calcium | 2 months
  Serum concentrations of calcium (mg/dL)
Iron | 2 months
  Serum concentrations of iron (mg/dL)
Sodium | 2 months
  Serum concentrations of sodium (mEq/L)
Potassium | 2 months
  Serum concentrations of potassium (mEq/L)
Phosphorus | 2 months
  Serum concentrations of phosphorus(mg/dL)
Folic acid | 2 months
  Serum concentrations of folic acid (ng/mL)
Vitamin B12 | 2 months
  Serum concentrations of vitamin B12 (pg/mL)
Vitamin D | 2 months
  Serum concentrations of vitamin D (ng/dL)
Body weight | 2 months
  Body weight (kg)
Waist circumference | 2 months
  Waist circumference (cm)
Body mass index | 2 months
  Body mass index (kg/m²)
Brain-derived neurotrophic factor (BDNF) | 2 months
  Plasma Brain-derived neurotrophic factor (ng or pg/mL)
Cortisol | 2 months
  Plasma cortisol (ug/dL)
Leptin | 2 months
  Plasma leptin (ng/mL)
Ghrelin | 2 months
  Plasma ghrelin (pg/mL)
Adrenocorticotropic Hormone (ACTH) | 2 months
  Plasma Adrenocorticotropic Hormone (pg/mL)
Hepcidin | 2 months
  Hepcidin (ng/mL)
Parathormone (PTH) | 2 months
  Parathormone (ng/mL)
Thyroid-Stimulating Hormone (TSH) | 2 months
  Thyroid-Stimulating Hormone (µIU/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Erasmo Trindade, PhD, Study Director — Federal University of Santa Catarina
Locations (1):
- Polydoro Ernani de São Thiago University Hospital, Florianópolis, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: Undecided